CLINICAL TRIAL: NCT03416777
Title: Faecal Microbiome as Determinant of the Effect of Diet on Colorectal-cancer Risk: Comparison of Meat Based Versus Pesco-vegetarian Diets (MeaTIc)
Brief Title: Meat-based Versus Pesco-vegetarian Diet and Colorectal Cancer
Acronym: MeaTIc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Francesco Sofi, Associate Professor of Clinical Nutrition, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MeaTIC-INTIMIC
Record Dates: First submitted 2018-01-08; First posted 2018-01-31 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Nutrition Aspect of Cancer; Diet Modification; Cancer of Colon
Keywords: vegetarian; meat; fish
MeSH Terms: conditions — Colonic Neoplasms | interventions — alpha-Tocopherol

STUDY DESIGN:
Intervention Model Description: Randomized parallel open dietary intervention study with 3 arms of intervention
Masking Description: In this trial blinding of participants and investigators will not be possible because of obvious differences between the intervention diets
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meat-based diet (MBD) (Active Comparator): Behavioral intervention with diet including 4 servings per week of red meat, 3 servings per week of processed meat, and 1 servings per week of poultry, for a total amount of 900 g per week of meat.
  Interventions: Behavioral: Meat-based diet
- Meat-based alpha-tocopherol (MBD-T) (Experimental): Behavioral intervention including diet with 4 servings per week of red meat, 3 servings per week of processed meat, and 1 servings per week of poultry, for a total amount of 900 g per week of meat with a dietary supplement of 100 mg/day of alpha-tocopherol in the form of tablet
  Interventions: Dietary Supplement: Meat-based diet supplemented with alpha-tocopherol (MBD-T)
- Pesco-vegetarian (PVD) (Experimental): Behavioral intervention with diet excluding fresh and processed meat, poultry but including 3 servings per week of any type of fish, excluding shellfish
  Interventions: Behavioral: Pesco-vegetarian diet

INTERVENTIONS:
Behavioral: Meat-based diet — Diet including 4 servings per week of red meat (1 serving = 150 g), 3 servings per week of processed meat (1 serving = 50 g), and 1 servings per week of poultry (1 serving = 150 g), for a total amount of 900 g per week of meat.
  Other Names: MBD
  Arms: Meat-based diet (MBD)
Dietary Supplement: Meat-based diet supplemented with alpha-tocopherol (MBD-T) — Dietary intervention like the MBD with supplementation of alpha-tocopherol at a dosage of 100 mg/die. Available evidence suggests that alpha-tocopherol may help prevent colon cancer by decreasing the formation of mutagens arising from the oxidation of faecal lipids, by decreasing oxidative stress in the epithelial cells of the colon and by molecular mechanisms that influence cell death, cell cycle and transcriptional events (Pierre 2013, Bastide 2016, Bastide 2017, Diallo 2016). It is important to note that 200 mg/day of tocopherol was administered to 20,000 women for 10 years without side effects (Lee et al.,2005).
  Other Names: MBD-T
  Arms: Meat-based alpha-tocopherol (MBD-T)
Behavioral: Pesco-vegetarian diet — Diet excluding fresh and processed meat, poultry but including 3 servings per week of any type of fish, excluding shellfish (1 serving = 150 g), for a total amount of 450 g per week. Diet will contain other sources of proteins (e.g. eggs, dairy, legumes/beans). There is suggestive evidence that fish and vegetable consumption has protective effects against CRC (Vieira et al., 2017).
  Other Names: PVD
  Arms: Pesco-vegetarian (PVD)

SUMMARY:
Colorectal cancer (CRC) is strongly affected by diet, with red and processed meat increasing risk. To understand the role of microbiome in this phenomenon and to identify specific microbiome/metabolomics profiles associated with CRC risk, will be studied: 1) healthy volunteers fed for 3 months with: a high-CRC risk diet (meat-based MBD), a normalized CRC risk diet (MBD plus alpha-tocopherol, MBD-T), a low-CRC risk diet (pesco-vegetarian, PVD). At the beginning and at the end of the intervention, gut microbiome profiles (metagenomics and metabolomics), and CRC biomarkers (genotoxicity, cytotoxicity, peroxidation in faecal water; lipid/glycemic indexes, inflammatory cytokines, oxidative stress), 2) Colon carcinogenesis: the same diets will be fed (3 months) to carcinogen-induced rats or to Pirc rats, mutated in Apc, the key gene in CRC; faecal microbiome profiles, will be correlated to carcinogenesis measuring preneoplastic lesions, colon tumours, and faecal and blood CRC biomarkers as in humans; 3) To further elucidate the mechanisms underlying the effect of different microbiomes in determining CRC risk, faeces from rats fed the experimental diets will be transplanted into carcinogen-induced germ-free rats, measuring how microbiome changes correlate with metabolome and disease outcomes. The results will provide fundamental insight in the role of microbiome in determining the effect of the diet, in particular red/processed meat intake, on CRC risk

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second leading cause of cancer death in Europe. The geographical variation of incidence demonstrates how environmental factors, chiefly dietary habits, play a major role in this disease. Convincing evidence suggests that risk of CRC is increased by red meat and processed meat consumption (classified, as regard cancer hazard as 2A and 1, respectively, WHO) and decreased by foods containing dietary fibers. As regarding other food groups, like fish, although epidemiological studies suggest a reduction of CRC risk associated with its consumption, the evidence for this link is considered limited; similarly, for non-starchy vegetables and fruits, although there is suggestive evidence of a protective effect, this is considered limited, and thus less convincing than that for red and processed meat.

Several hypotheses are proposed to explain the positive association between red, processed meat and CRC: meat-based diets contain mutagens-carcinogens formed during cooking, but also lipid peroxidation and N-nitroso compounds whose formation is catalyzed by heme in the colon. Accordingly, recent experimental and epidemiological studies on the E3N cohort and on the randomized placebo-controlled trial SUVIMAX carried out by our group, demonstrated the central role of heme iron in the positive association between meat and CRC. According to these studies, this effect is largely explained by the ability of heme iron to catalyze peroxidation and induce high luminal polyunsaturated fatty acids (PUFAs) peroxidation, forming cytotoxic and genotoxic alkenals which will in turn induce positive selection of precancerous cells mutated for Apc, the key gene in CRC. On this basis, it was also demonstrated that antioxidants, in particular tocopherol, modulate the risk of cancer associated with red meat in experimental animals and humans by controlling heme iron-induced peroxidation. Recent data from the investigators demonstrated that microbiota is involved in the heme-induced peroxidation and it has been reported that the gut microbiota is required for heme-induced epithelial hyperproliferation and hyperplasia because of the capacity to reduce mucus barrier function. Notwithstanding these reports, the role of gut microbiome in determining cancer risk associated with red and processed meat is not clear.

Microbial fermentation of plant-based foods, associated with a low CRC risk increases intestinal Short Chain Fatty Acids (SCFAs), among which butyrate, endowed with antineoplastic activity through its inhibition of histone deacetylase and promotion of apoptosis and microbial activated phytochemicals, such as polyphenols with anti-inflammatory and antioxidant activities. Accordingly, it is also known that the process of fermenting fibers to SCFAs needs intestinal bacteria because germ-free mice produce almost no SCFAs. These data clearly indicate that, at least part of the effect of the diet on colon carcinogenesis is mediated by the intestinal microbiome. Accordingly, it is well know that diet shapes gut microbiome composition, as described in a human rural population study and emerging evidences implicate an involvement of the gut microbiota in CRC. Microorganisms and their metabolites have been proposed to promote carcinogenesis by several mechanisms, including induction of inflammatory signaling pathways, genetic mutations, and epigenetic dysregulation. Recently, a review conducted on 31 studies (human and animal models) has shown that certain bacterial groups are increased (eg. Fusobacterium spp, Alistipes, Staphylococcaceae, Akkermansia spp. and Methanobacteriales), while others (eg. Bifidobacterium, Lactobacillus, Faecalibacterium spp) are consistently diminished in CRC, with consequent increase of potentially carcinogenic metabolites (nitrogen compounds, bile acids) and decrease of SCFAs (eg. butyrate). However, it is still not clear whether dysbiosis (imbalanced microbiota) is the cause or consequence of CRC. Tumorigenesis can indeed produce inflammation, ulceration and necrosis of the mucosa, by changing the microenvironment and growth conditions for different microorganisms, thus it is difficult to understand what comes first. And furthermore, how dietary risk is mediated by the interaction with the gut microbiome? How can the modulation of the microbiome promote or prevent the development of a microenvironment containing pro-inflammatory and carcinogenic metabolites that favour the neoplastic initiation process? Cohort studies with subjects consuming various types of diets (i.e omnivores, vegetarians, vegans) suggest that diet alters the intestinal microbiome as well as the cytotoxic and genotoxic activities of the luminal colonic content. In a study on ten volunteers following for 5 days a strictly vegetarian diet and then moving to a strictly carnivorous diet, it was demonstrated that the intestinal bacteria react very quickly (24-48 hours). In particular, bacterial species capable of digesting complex carbohydrates prevailed during the vegetarian diet period while during the animal proteins based diet, specific bacterial species were selected, such as Bilophila wadsworthia, which are able to metabolize proteins and produce toxic compounds like secondary bile acids (BA, promoters of carcinogenesis) and with great pro-inflammatory potential. Feeding a high-fibre low-fat African-style diet to African Americans at high risk of colon cancer and, vice versa, feeding a high-fat, low-fiber western style diet to rural Africans at low risk of cancer, causes variation in microbiome and in parameters associated with CRC risk. Preliminary data in humans also demonstrate that when an animal-based diet rich in fat and simple sugars is introduced into a traditional African diet, composed of cereals, legumes and vegetables, the gut microbiome shifts, leading to progressive loss of biochemical functions associated with SCFAs production, suggesting indeed that faecal microbiome may act as determinant of colon cancer risk related to the diet. Regarding heme iron, the investigators recently demonstrated that after a short term exposure (14 days), the gut microbiota of heme-fed rats was enriched with Enterobacteriaceae and B. fragilis whereas Roseburia spp. and Lactobacillus spp. were underrepresented. Notably, Enterobacteriaceae expansion is also found in Inflammatory Bowel Disease (IBD) patients at high risk for CRC and can induce inflammation in the host gut epithelium. Moreover, B. fragilis has been associated with inflammation-induced colon cancer. It has also been shown that Lactobacilli can inhibit iron-induced lipoperoxidation. Remarkably, the gut microbiota modulations observed after heme iron intake present similarities with that observed comparing colorectal cancer patients and healthy volunteers. However, although the association between gut microbiota and CRC is conceptually interesting, these outcomes do not help to explain the mechanism behind the modulations of the gut microbiota by the diet and the consequent impact on CRC risk. In addition, while many studies have been conducted for bacteria, fungi have been virtually unexplored by metagenomic studies, yet they are emerging as key players involved in autoimmune or inflammatory disorders, as recently demonstrated. Their relative under-representation in number compared to bacteria, results in their underestimation, since fungal DNA often cannot be purified using standard approaches. Preliminary results revealed a higher frequency of S. cerevisiae in IBD, a group pathologies associated with increased risk of CRC.

ELIGIBILITY:
Inclusion Criteria:

* clinically healthy (both sexes)
* age >18 years and ≤ 50 years.

The study population will be selected with an age ranging from 18 to 50 years because after 50 years the risk for CRC shows a significant increase in incidence. In fact, more than 90% of the people diagnosed with the disease are older than 50, with the average age at the time of diagnosis being 64 (Amersi et al., 2005). With respect to gender, its role in the development of colorectal cancer remains unclear (Amersi et al., 2005).

Exclusion Criteria:

* Presence of current illness or unstable conditions
* Current or recent (past 2 months) use of antibiotics or probiotics
* Pregnancy or intention to become pregnant in the next 12 months or lactation
* Current smoking habit
* Current or recent (past 2 months) adoption of a vegetarian diet

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
DNA damage | 3 months
  Decrease (<25%) of DNA damage by faecal water (genotoxicity), using comet assay in a cellular model

SECONDARY OUTCOMES:
Microbiome and metabolomics profiles | 3 months
  Changes of microbiome and the relative metabolomics profiles from baseline
Peroxidation | 3 months
  Global and specific peroxidation of omega-3 and omega-6 of the faecal water change from baseline
Inflammatory parameters | 3 months
  Pro- and anti-inflammatory profile's change from baseline
Oxidative stress | 3 months
  Oxidative stress profile's change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Casini, MD, Study Director — University of Florence
Locations (1):
- Unit of Clinical Nutrition, University Hospital of Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Femia AP, Luceri C, Soares PV, Lodovici M, Caderni G. Multiple mucin depleted foci, high proliferation and low apoptotic response in the onset of colon carcinogenesis of the PIRC rat, mutated in Apc. Int J Cancer. 2015 Mar 15;136(6):E488-95. doi: 10.1002/ijc.29232. Epub 2014 Oct 6. PMID 25257656
- [Background] Bastide NM, Naud N, Nassy G, Vendeuvre JL, Tache S, Gueraud F, Hobbs DA, Kuhnle GG, Corpet DE, Pierre FH. Red Wine and Pomegranate Extracts Suppress Cured Meat Promotion of Colonic Mucin-Depleted Foci in Carcinogen-Induced Rats. Nutr Cancer. 2017 Feb-Mar;69(2):289-298. doi: 10.1080/01635581.2017.1263745. Epub 2017 Jan 17. PMID 28094544
- [Background] Caderni G, Femia AP, Giannini A, Favuzza A, Luceri C, Salvadori M, Dolara P. Identification of mucin-depleted foci in the unsectioned colon of azoxymethane-treated rats: correlation with carcinogenesis. Cancer Res. 2003 May 15;63(10):2388-92. PMID 12750256
- [Background] Irrazabal T, Belcheva A, Girardin SE, Martin A, Philpott DJ. The multifaceted role of the intestinal microbiota in colon cancer. Mol Cell. 2014 Apr 24;54(2):309-20. doi: 10.1016/j.molcel.2014.03.039. PMID 24766895
- [Background] Pierre F, Peiro G, Tache S, Cross AJ, Bingham SA, Gasc N, Gottardi G, Corpet DE, Gueraud F. New marker of colon cancer risk associated with heme intake: 1,4-dihydroxynonane mercapturic acid. Cancer Epidemiol Biomarkers Prev. 2006 Nov;15(11):2274-9. doi: 10.1158/1055-9965.EPI-06-0085. PMID 17119057
- [Background] Gueraud F, Tache S, Steghens JP, Milkovic L, Borovic-Sunjic S, Zarkovic N, Gaultier E, Naud N, Helies-Toussaint C, Pierre F, Priymenko N. Dietary polyunsaturated fatty acids and heme iron induce oxidative stress biomarkers and a cancer promoting environment in the colon of rats. Free Radic Biol Med. 2015 Jun;83:192-200. doi: 10.1016/j.freeradbiomed.2015.02.023. Epub 2015 Mar 3. PMID 25744414
- [Background] De Filippis F, Pellegrini N, Vannini L, Jeffery IB, La Storia A, Laghi L, Serrazanetti DI, Di Cagno R, Ferrocino I, Lazzi C, Turroni S, Cocolin L, Brigidi P, Neviani E, Gobbetti M, O'Toole PW, Ercolini D. High-level adherence to a Mediterranean diet beneficially impacts the gut microbiota and associated metabolome. Gut. 2016 Nov;65(11):1812-1821. doi: 10.1136/gutjnl-2015-309957. Epub 2015 Sep 28. PMID 26416813
- [Result] De Filippo C, Cavalieri D, Di Paola M, Ramazzotti M, Poullet JB, Massart S, Collini S, Pieraccini G, Lionetti P. Impact of diet in shaping gut microbiota revealed by a comparative study in children from Europe and rural Africa. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14691-6. doi: 10.1073/pnas.1005963107. Epub 2010 Aug 2. PMID 20679230
- [Result] Albanese D, De Filippo C, Cavalieri D, Donati C. Explaining diversity in metagenomic datasets by phylogenetic-based feature weighting. PLoS Comput Biol. 2015 Mar 27;11(3):e1004186. doi: 10.1371/journal.pcbi.1004186. eCollection 2015 Mar. PMID 25815895
- [Result] Pierre FH, Martin OC, Santarelli RL, Tache S, Naud N, Gueraud F, Audebert M, Dupuy J, Meunier N, Attaix D, Vendeuvre JL, Mirvish SS, Kuhnle GC, Cano N, Corpet DE. Calcium and alpha-tocopherol suppress cured-meat promotion of chemically induced colon carcinogenesis in rats and reduce associated biomarkers in human volunteers. Am J Clin Nutr. 2013 Nov;98(5):1255-62. doi: 10.3945/ajcn.113.061069. Epub 2013 Sep 11. PMID 24025632
- [Derived] Dinu M, Ristori S, Pagliai G, Lotti S, Meriggi N, Nerini A, Chevolleau S, Bowman J, Caderni G, Colombini B, Gerard P, Giovannelli L, Gueraud F, Marcucci R, Pierre F, De Filippo C, Sofi F. Effects of meat-based, meat-based with alpha-tocopherol, and pesco-vegetarian diets on biomarkers associated with colorectal cancer risk: a randomized behavioral intervention trial. Sci Rep. 2025 Dec 8;16(1):1502. doi: 10.1038/s41598-025-31410-6. PMID 41361349
- [Derived] Sofi F, Dinu M, Pagliai G, Pierre F, Gueraud F, Bowman J, Gerard P, Longo V, Giovannelli L, Caderni G, de Filippo C. Fecal microbiome as determinant of the effect of diet on colorectal cancer risk: comparison of meat-based versus pesco-vegetarian diets (the MeaTIc study). Trials. 2019 Dec 9;20(1):688. doi: 10.1186/s13063-019-3801-x. PMID 31815647